CLINICAL TRIAL: NCT05106985
Title: A Single Case Experimental Design Study of a Reminder App for Supporting Adherence to Personalised Treatment Goals in Parkinson's Disease
Brief Title: A Reminder App for Supporting Adherence to Treatment Goals in Parkinson's Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NHS Greater Glasgow and Clyde (Other)
Collaborators: University of Glasgow (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Supportive Care
Other Study IDs: GN21NE440
Record Dates: First submitted 2021-10-25; First posted 2021-11-04 (Actual); Last update posted 2022-09-26 (Actual); Status verified 2022-09

CONDITIONS: Parkinson Disease
Keywords: Parkinson's disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Intervention Model Description: Single case experimental design: Multiple Baseline Design
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ApplTree Reminder app (Experimental): Following a randomised baseline period, each participant will use the ApplTree reminder app for 22 days to support adherence to goal-related tasks
  Interventions: Device: ApplTree reminder app

INTERVENTIONS:
Device: ApplTree reminder app — The reminder app will be introduced to participants to support adherence to chosen goal-related tasks. Reminder app will be introduced following a baseline phase of 10, 16 or 22 days. The duration of the baseline phase will be randomly assigned using an online random number generator.

SUMMARY:
Parkinson's Disease is a progressive condition which affects the nervous system causing tremors, slowed movement and often causes problems with memory and initiation. Treatment management can be complex and challenging for patients and families. Poor memory in Parkinson's disease has been shown to reduce a person's ability to manage activities of daily living, including tasks associated with treatment such a taking medications. However, patients with Parkinson's have been shown to benefit from external reminders.

The aim of this research project is to investigate whether the use of a reminder app that has been designed for use by people with cognitive difficulties improves completion of activities related to therapy goals in people with Parkinson's Disease, aiding self-management of their condition.

Patients seen in movement disorder clinics in NHS Greater Glasgow and Clyde with a diagnosis of Parkinson's disease, and a partner or carer who can monitor progress, will be invited to participate. Measures of memory, emotional wellbeing and quality of life will be completed to characterise each participant. Participants will have a randomly allocated initial baseline period of either 10, 16 or 22 days in which their rate of completion of intended activities will be monitored. Then, during the intervention period of 3 weeks (21 days) the ApplTree app will be introduced to remind participants of treatment goals. Participants will create specific and personalised treatment goals at the beginning of the monitoring period. Goals will be everyday activities relevant to the management and treatment of Parkinson's disease. The number of goals is not limited and will depend on how frequent targeted behaviours are. However, at least one target behaviour a day in total will be recommended. E.g. Completing daily exercises. Partners will monitor their goal attainment, via a daily/weekly monitoring form in both phases of the study.

DETAILED DESCRIPTION:
Aims:

The aim of this project is to investigate whether the use of a recently developed reminder app ApplTree improves attainment of personalised specific treatment goals in people with Parkinson's disease (PD).

Hypothesis:

The hypothesis of this study is that introduction of the reminder app will significantly improve attainment of treatment goals.

Methods

Design:

A single case experimental design (SCED) will be utilised with multiple baselines across participants with randomisation of the onset of the intervention phase for each participant.

Participants:

Participants will have a clinical diagnosis of PD. Further, the Parkinson's care team or the individual will have expressed concerns about adherence or attainment of treatment goals. Due to the design of the study, participants will be required to own a smart phone and have a partner or significant other who is able to, and consents to, monitor and support the participant's goal attainment as the nominated person.

Recruitment:

PD patients will be recruited via the movement disorder teams and movement disorder neurology clinics in Greater Glasgow and Clyde NHS Trust (GGC) via their Parkinson's consultant, named Parkinson's nurse specialist, occupational therapist, or physiotherapist within the team.

Measures:

Pre intervention measures:

All measures are validated for PD and recommended by the Movement Disorder Society (MDS).

* A cognitive screen will be completed with all participants, the Montreal Cognitive Assessment.
* Parkinson's Disease Quality of Life Questionnaire. A proxy-rating version will also be utilised.
* Prospective and Retrospective Memory Questionnaire (PRMQ). A proxy-rating version of the PRMQ will also be utilised to alleviate limitations of self-report measures and build a broader picture.
* Apathy Scale (AS).
* Currently, no measure of anxiety is recommended by the MDS, therefore, the Generalised Anxiety Disorder severity index (GAD-7) and the Patient Health Questionnaire (PHQ-9) will be used to assess emotional wellbeing.

A weekly/daily monitoring form will be used by the partner during all phases of the intervention to record completion of intended goal related tasks (e.g., taking medication on time, completing prescribed exercises, nutritional snack, attending support group).

Procedure:

The study will run in batches of three participants, with replication of the design across the second set of three. The data collection phase for each participant will vary based on completing at least 5 data points within both the baseline and intervention phase and will range from 31-43 days for each participant. It is hoped that the timeframes for goals will require at least one reminder activity per day and so a two-day period will represent one datapoint. Participants will be assigned to a baseline period of 10, 16 or 22 days and an intervention period of 21 days (3 weeks).

Schedule:

1. Members of the movement disorder teams in GGC will be asked to review caseloads for suitable participants, based on inclusion and exclusion criteria. Participants will have a diagnosis of Parkinson's disease, have a consenting partner or carer, have use of a mobile phone and have difficulty adhering to treatment goals.
2. Potential participants and their carers/partners (nominated person) will be sent out the participant information sheet by post or be given them by a member of their clinical team during a clinic appointment. Potential participants will be able to indicate their willingness to discuss participation in the research with the researcher by returning a consent to be contacted form by pre-post to the researcher directly or by emailing the researcher informing them of their agreement for contact.
3. Alternatively in cases where participant information is given in the appointment, participants can inform the clinical team member at their clinic appointment of their agreement for contact. In this instance staff will then send contact details of potential participants who have agreed for contact along to the researcher, via NHS secure email.
4. Participants and nominated persons who consent to contact will be given a phone call to discuss the study in more detail and have the opportunity to ask any questions and, if ready, make a decision on whether they would like to participate and if undecided will be given a follow up call in 2 -5 days (depending on when is convenient for them). Inclusion and exclusion criteria will also be reviewed at this point to ensure eligibility.
5. Eligible participants and nominated persons will then meet with the researcher initially to complete written consent form and pre intervention measures. This meeting will be either face-to-face in an NHS building, face-to-face in their own home or via video call, depending on participant preferences and travel limitations.
6. Participants and nominated persons will then meet with the researcher a second time (Face-to-face or Video call) to discuss and formulate specific and personalised treatment/therapy goals. Discussion of goals will be informed by pre-intervention measures, partners and participants own views. Goals will be relevant to the management and treatment of Parkinson's Disease and have a memory and motivational component such as reminders for medication regime or physical exercises.
7. A weekly monitoring form will then be given to participants' nominated person to record completion of intended goal related tasks (e.g., taking medication on time, completing prescribed exercises, nutritional snack, attending support group) and the baseline phase will begin for a duration of 10, 16 or 22 days the following day. The duration of the baseline phase will be randomly assigned using an online random number generator.
8. The nominated person will receive a weekly reminder call to ensure the weekly monitoring form is being completed and to troubleshoot any problems.
9. The nominated person will receive a reminder text on a daily basis to ensure the form is being completed daily.
10. At the end of the baseline phase, participants and partners will meet with the researcher (Face to face or video call) to receive a training session on using the app and to input reminders for specific goal related actions.
11. Participants will then start an intervention phase of 22 days and partners will continue to use the monitoring form provided.
12. Participants will receive a weekly phone call to troubleshoot any problems.
13. The nominated person will receive a reminder text on a daily basis to ensure the monitoring form is completed daily.
14. At the end of the intervention stage participants and nominated persons will meet with the researcher a final time for a debrief (face-to-face or video call).

Setting:

Meetings with participants will be in an agreed NHS building, remote video call via attend anywhere, or in some cases in the participants own home. Due to the nature of health conditions and travel limitations within the population, the preferences of the participant and their nominated person will be given priority for arranging meetings. Current Scottish government/NHS GG&C guidance surrounding COVID-19 will also be taken into account. Telephone calls and video calls will be completed by the researcher from an NHS premises, to ensure confidentiality of data collected.

Materials:

ApplTree is a reminding app designed to be used by people with cognitive impairments as a result of acquired brain injury. ApplTree has a narrow/deep user interface design which presents a small amount of information at a time to minimise the burden on people with cognitive impairment. Each participant will download the ApplTree app onto their own smart device. The app is free to use and maintained by Glasgow University Software Services (GUSS).

Analysis Plan:

The primary outcome measure will be the percentage of goal related tasks carried out independently (i.e., without prompting from another person) per two-day period. The primary outcome is measured via the daily monitoring form, completed by participant's nominated person. In line with recommendations for analysis of SCED data, the data will be analysed through visual analysis of graphs and Tau-U analysis to determine whether a significant improvement is found between baseline and intervention phase.

Sample Size:

The Risk of Bias in N of 1 Trials (RoBiNT) recommends that SCED designs provide at least three demonstrations of the treatment effect. In a multiple baseline across participants design this means a minimum of three participants. Additionally, the RoBiNT highlights the importance of replication, referring to replication of the overall study, meaning replication of the set of three participants. Hence, the present study will aim to recruit a minimum of six participants, and to allow for possible withdrawals the aim will be to recruit nine participants.

ELIGIBILITY:
Inclusion Criteria:

* A clinical diagnosis of PD.
* Participants will be required to own a smart phone
* Have a partner or significant other who is able to, and consents to, monitor and support the participant's goal attainment through daily monitoring forms.
* Possible concerns around adherence or attainment of treatment goals by Movement disorder team, patient or significant other

Exclusion Criteria:

* A diagnosis of dementia
* Pre-existing neurological or severe and enduring psychiatric disorder.
* Do not own a smart phone capable of downloading apps.
* Sensory deficits preventing the use of a smart device/phone.
* Are currently involved in any other research study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2022-01-20 (Actual); Primary Completion 2022-07-30 (Actual); Study Completion 2022-09-02 (Actual)

PRIMARY OUTCOMES:
Goal-related tasks completed | 22 days
  The primary outcome measure will be the percentage of goal related tasks carried out independently (i.e., without prompting from another person) per two-day period. The primary outcome is measured via the daily monitoring form, completed by participant's nominated person.

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Evans, Principal Investigator — University of Glasgow
Locations (1):
- NHS Greater Glasgow and Clyde, Glasgow, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
It is standard practice in reporting SCED studies to provide raw data for each participant within the study write up. This means that data are available for future researchers (e.g. for the purpose of meta-analysis). Care will be taken to ensure included data ensures anonymity of participants and that demographic information is kept to a minimum so that they cannot be identified from the data.
Supporting Information: CSR
Time Frame: Upon publication
Access Criteria: Individual patient date are routinely reported in study outputs from Single Case Experimental Design studies, in line with methodological and reporting quality guidelines.

REFERENCES:
- [Background] Jamieson M, Cullen B, Lennon M, Brewster S, Evans J. Designing ApplTree: usable scheduling software for people with cognitive impairments. Disabil Rehabil Assist Technol. 2022 Apr;17(3):338-348. doi: 10.1080/17483107.2020.1785560. Epub 2020 Jul 7. PMID 32633592
- [Background] Tate RL, Perdices M, Rosenkoetter U, Wakim D, Godbee K, Togher L, McDonald S. Revision of a method quality rating scale for single-case experimental designs and n-of-1 trials: the 15-item Risk of Bias in N-of-1 Trials (RoBiNT) Scale. Neuropsychol Rehabil. 2013;23(5):619-38. doi: 10.1080/09602011.2013.824383. Epub 2013 Sep 9. PMID 24050810
- [Background] Parker RI, Vannest KJ, Davis JL, Sauber SB. Combining nonoverlap and trend for single-case research: Tau-U. Behav Ther. 2011 Jun;42(2):284-99. doi: 10.1016/j.beth.2010.08.006. Epub 2011 Feb 3. PMID 21496513
- [Background] Spitzer RL, Kroenke K, Williams JB, Lowe B. A brief measure for assessing generalized anxiety disorder: the GAD-7. Arch Intern Med. 2006 May 22;166(10):1092-7. doi: 10.1001/archinte.166.10.1092. PMID 16717171
- [Background] Starkstein SE, Mayberg HS, Preziosi TJ, Andrezejewski P, Leiguarda R, Robinson RG. Reliability, validity, and clinical correlates of apathy in Parkinson's disease. J Neuropsychiatry Clin Neurosci. 1992 Spring;4(2):134-9. doi: 10.1176/jnp.4.2.134. PMID 1627973
- [Background] Spitzer RL, Kroenke K, Williams JB. Validation and utility of a self-report version of PRIME-MD: the PHQ primary care study. Primary Care Evaluation of Mental Disorders. Patient Health Questionnaire. JAMA. 1999 Nov 10;282(18):1737-44. doi: 10.1001/jama.282.18.1737. PMID 10568646
- [Background] Peto V, Jenkinson C, Fitzpatrick R. PDQ-39: a review of the development, validation and application of a Parkinson's disease quality of life questionnaire and its associated measures. J Neurol. 1998 May;245 Suppl 1:S10-4. doi: 10.1007/pl00007730. PMID 9617716
- [Background] Nasreddine ZS, Phillips NA, Bedirian V, Charbonneau S, Whitehead V, Collin I, Cummings JL, Chertkow H. The Montreal Cognitive Assessment, MoCA: a brief screening tool for mild cognitive impairment. J Am Geriatr Soc. 2005 Apr;53(4):695-9. doi: 10.1111/j.1532-5415.2005.53221.x. PMID 15817019